CLINICAL TRIAL: NCT06095973
Title: A Single Center, Single-blind, Randomized, Dose-escalation, Parallel, Placebo and Active-controlled, Single Dose, Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GB-6002 Local Infiltration in Healthy Male Adults
Brief Title: Dose-Escalation, Single Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GB-6002 Local Infiltration in Healthy Male Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: G2GBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GB6002101
Record Dates: First submitted 2023-10-04; First posted 2023-10-23 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: sequential
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort B (Other): Experimental : GB-6002 for subcutaneous injection at intermediate A dose. Placebo Comparator: Placebo for subcutaneous injection at intermediate intermediate A dose.
  Active Comparator: Naropin injection(Ropivacaine hydrochloride), single dose.
  Interventions: Drug: GB-6002; Drug: Placebo; Drug: Naropin injection
- Cohort C (Other): Experimental : GB-6002 for subcutaneous injection at intermediate B dose. Placebo Comparator: Placebo for subcutaneous injection at intermediate B dose. Active Comparator: Naropin injection(Ropivacaine hydrochloride), single dose.
  Interventions: Drug: GB-6002; Drug: Placebo; Drug: Naropin injection
- Cohort D (Other): Experimental : GB-6002 for subcutaneous injection at high dose. Placebo Comparator: Placebo for subcutaneous injection at high dose. Active Comparator: Naropin injection(Ropivacaine hydrochloride), single dose.
  Interventions: Drug: GB-6002; Drug: Placebo; Drug: Naropin injection
- Cohort A (Other): Experimental : GB-6002 for subcutaneous injection at low dose. Placebo Comparator: Placebo for subcutaneous injection at low dose. Active Comparator: Naropin injection(Ropivacaine hydrochloride), single dose.
  Interventions: Drug: GB-6002; Drug: Placebo; Drug: Naropin injection

INTERVENTIONS:
Drug: GB-6002 — Depending on the cohort, volume will be varied to administer.
Drug: Placebo — Depending on the cohort, volume will be varied to administer. Volume to be matched with the active investigational drug in the respective cohort.
Drug: Naropin injection — Single dose of Naropin s.c. injection.

SUMMARY:
This study is to evaluate the safety and tolerability of single dose of GB-6002 (Ropivacaine) Local Infiltration in healthy male Adults. And, It is to compare pharmacokinetic characteristics of GB-6002 single dose injection with active comparator.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males,19 to 55 years of age, inclusive at the time of screening visit.
* At the time of screening, those with a body weight of 55 kg or more and a BMI (Body Mass Index) within 18.0 to 27.0 kg/m², inclusive.
* Subjects who do not have plans to receive COVID-19(coronavirus disease 2019) vaccination during the clinical trial starting from 14 days prior to the first administration of investigational drug.
* Subjects who have understood the purpose of this clinical trial, voluntarily chosen to participate, and provided written consent to adhere to the restrictions.

Exclusion Criteria:

* Subjects with clinically significant cardiovascular, respiratory, hepatic, renal, neurological, endocrine, hematologic, oncological, psychiatric, or urological conditions, or a history related to such conditions.
* Subjects with systolic blood pressure less than 90 mmHg or greater than 150 mmHg, or diastolic blood pressure less than 50 mmHg or greater than 100 mmHg during the screening assessments.
* Subjects who exhibited clinically significant abnormalities in physical examination, clinical laboratory tests, or electrocardiograms during the screening assessments.
* Subjects known to be hypersensitive to Investigational Product and its components.
* Subjects who have continued to drink alcohol within 1 month prior to the first administration of Investigational Product or who are unable to abstain from alcohol during the clinical trial.
* Subjects who smoked continuously within 1 month prior to the first administration of Investigational Product or are unable to quit smoking during the clinical trial.
* Subjects who has taken drugs that induce or inhibit drug metabolism enzymes, such as barbiturates, within 1 month prior to the first administration of Investigational Product.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Day 1 to Day 14
  Number of subjects and Incidences with adverse events by Study arm. Number of subjects and Incidences with Injection site assessments for nodules by Study arm.
Clinical Laboratory tests | Day 1 to Day 14
  Incidence of abnormal clinically significant clinical laboratory test results (Hematology, Blood Chemistry Test, Urine Test, Blood Coagulation Test, Serum Test and Urine Drug Screening Test, etc) by study arm.
Physical examination | Day 1 to Day 14
  Incidence of abnormal clinically significant Physical examination results by Study arm.
Vital signs | Day 1 to Day 14
  Incidence of abnormal clinically significant vital signs(Systolic and Diastolic Blood Pressure, Pulse Rate, Body Temperature) results by Study arm.
Electrocardiograms | Day 1 to Day 14
  Incidence of abnormal clinically significant ECG results by Study arm.

SECONDARY OUTCOMES:
Pharmacokinetics(Cmax) | Day 1 to Day 14
Pharmacokinetics(AUCt) | Day 1 to Day 14
Pharmacokinetics(AUCinf) | Day 1 to Day 14
Pharmacokinetics(Tmax) | Day 1 to Day 14
Pharmacokinetics(t1/2) | Day 1 to Day 14
Pharmacokinetics(CL/F) | Day 1 to Day 14
Pharmacokinetics(Vz/F) | Day 1 to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Yoon, Principal Investigator — Republic of Korea, Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea